CLINICAL TRIAL: NCT03424161
Title: Multi-Center, Clinical Evaluation of the Cutera Secret RF Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cutera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C-18-SRF01
Record Dates: First submitted 2018-01-25; First posted 2018-02-06 (Actual); Results first posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Skin Quality

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Secret RF (Other): Treatment with Secret RF for skin quality
  Interventions: Device: Secret RF

INTERVENTIONS:
Device: Secret RF — Subjects will receive treatment with the Secret RF device

SUMMARY:
The objectives of this study are to evaluate the efficacy and safety of the Cutera Secret RF device.

DETAILED DESCRIPTION:
This is a multi-center, study in approximately 40 subjects, ages 18 and older. Subjects will receive treatments and will be followed at 4 and 12 weeks post the final treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be able to read, understand and sign the Informed Consent Form.
2. Female or Male, age 18 and older
3. Willing to undergo treatments with Secret RF.
4. Willing to have very limited sun exposure and use sunscreen on the treatment area every day for the duration of the study, including the follow-up period.
5. Subject must adhere to the follow-up schedule and study instructions.
6. Agree to not undergo any other cosmetic procedure(s) or treatment(s) on the treatment area during the study and has no intention of having such procedures performed during the course of the study.
7. Willing to have digital photographs taken of the treatment area and agree to use of photographs for presentation, (educational and/or marketing), publications, and any additional marketing purposes.
8. For female subjects: not pregnant or lactating and is either post-menopausal, surgically sterilized, or using a medically acceptable form of birth control prior to enrollment and during the entire course of the study.

Exclusion Criteria:

1. Participation in a clinical trial of another device or drug within 1 month of study participation, or during the study period.
2. History of clotting disorders and/or current use of blood thinning medications.
3. History of autoimmune disorders or diabetes.
4. Cardiac pacemaker or active implantable metal device in the treatment area.
5. Allergies to metals i.e. gold.
6. Has a history of squamous cell carcinoma or melanoma in the treatment area.
7. Significant uncontrolled concurrent illness that in the opinion of the Investigator would make the subject unsuitable for inclusion.
8. History of any disease or condition that could impair wound healing.
9. History of keloid formation or abnormal/delayed wound healing.
10. History of disease stimulated by heat, such as recurrent herpes simplex and/or herpes zoster (shingles) in the treatment area, unless treatment is conducted following a prophylactic regimen.
11. Use of topical agents one week prior to treatment that may cause facial sensitivity.
12. Suffering from significant skin conditions in the treated areas or inflammatory skin conditions, including but not limited to, open lacerations or abrasions, hidradenitis, rash, infection , or dermatitis of the treatment area prior to treatment (duration of resolution as per the Investigator's discretion).
13. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study or a condition that would compromise the subject's ability to comply with the study requirements.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2018-10-08 (Actual); Study Completion 2018-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Ronan, MD, Principal Investigator — Cutera Research Center
Locations (1):
- Cutera Research Center, Brisbane, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Secret RF
Started | 27
Completed | 10
Not Completed | 17

BASELINE CHARACTERISTICS:
Arm/Group | Secret RF
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Aesthetic Improvement
Description: Efficacy of treatment(s) with Cutera Secret RF measuring the global skin improvement at the 4 week follow-up visit, and at the 12 week follow-up visit as assessed by the study investigator using GAIS: Global Aesthetic Improvement Scale (+4=Very Significant Improvement, +3=Significant Improvement, +2=Moderate Improvement, +1=Mild Improvement, or 0=No Change Higher scores indicate better outcomes
Time Frame: at 4 weeks follow-up and 12 weeks follow-up
Population: 3 subjects has GAIS measurements available at both the 4 and 12 week follow ups 5 subjects had GAIS measurements only available at the 4 week follow up 2 subjects had GAIS measurements only available at the 12 week follow up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Secret RF
Number analyzed (Participants) | 10
score on a scale
  GAIS at the 4 week follow up: number analyzed (Participants) | 8
  GAIS at the 4 week follow up | 1.63 (0.92)
  GAIS at the 12 week follow up: number analyzed (Participants) | 5
  GAIS at the 12 week follow up | 2 (0.71)

ADVERSE EVENTS:
Time Frame: 12 weeks post final treatment, up to 8 months
Arm/Group | Secret RF
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 27/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Secret RF (N=27)
Edema (Skin and subcutaneous tissue disorders) | 27
Erythema (Skin and subcutaneous tissue disorders) | 27
Pain (Skin and subcutaneous tissue disorders) | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-03-29): https://cdn.clinicaltrials.gov/large-docs/61/NCT03424161/Prot_001.pdf